CLINICAL TRIAL: NCT04786782
Title: Clinical Management of Patients With Cirrhotic Portal Hypertension Based on the Noninvasive Portal Pressure Gradient (vPPG) Detecting Software, a Prospective and Controlled Cohort Study
Brief Title: The vPPG-detecting Software Guided Management of Cirrhotic Portal Hypertension
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Changqing Yang (Other)
Responsible Party: Sponsor-Investigator, Changqing Yang, Principal Investigator,Head of Gastroenterology and Hepatology, Chief Physician, Professor, Shanghai Tongji Hospital, Tongji University School of Medicine
Organization: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Other Study IDs: Yang-20210205
Record Dates: First submitted 2021-03-02; First posted 2021-03-08 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Portal Hypertension; Cirrhosis, Liver
Keywords: Virtual portal pressure gradient; Enhanced upper abdominal CT; Portal ultrasound; Portal hypertension; Cirrhosis
MeSH Terms: conditions — Hypertension, Portal; Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Three-dimensional reconstruction group: Portal hypertension is controlled with upper endoscopic screening and vPPG was detected by the noninvasive PPG-detecting software
  Interventions: Diagnostic Test: PPG-detecting software
- Natural follow-up group: Portal hypertension is controlled with the most updated guideline for clinical practice, namely, cirrhotic patients with either liver stiffness measurement >15kPa or PLT<150*10^9 should be screened with upper GI endoscopy and treated according to endoscopic results
  Interventions: Diagnostic Test: LSM and PLT count

INTERVENTIONS:
Diagnostic Test: PPG-detecting software — Virtual PPG (vPPG) of patients in experimental group is calculated based on anatomical and hemodynamic information of portal system collected by ultrasound and CT tests.
  Groups: Three-dimensional reconstruction group
Diagnostic Test: LSM and PLT count — Patients whose LSM >15kPa, or PLT count < 150*10^9 should be screened with upper GI endoscopy
  Groups: Natural follow-up group

SUMMARY:
The aim of this study is to investigate the possibilities and effectiveness of managing cirrhotic portal hypertension using the non-invasive portal pressure gradient (PPG) detecting software. In this study, the three-dimensional reconstruction and natural follow-up methods have been respectively applied in the experimental (1st) and active comparator (2nd) group. The virtual PPG is calculated with anatomical and hemodynamic information of portal system collected by ultrasound and CT tests. Cirrhosis patients in the 1st group, with calculated vPPG values, are managed with upper GI endoscopic results. Besides, patients in the 2nd group, are managed according to the most updated Chinese clinical guideline for cirrhotic portal hypertension, namely, patients with either liver stiffness measurement (LSM) >15kPa or PLT count <150*10^9 should be screened and treated with upper GI endoscopy. The morbidity of decompensated cirrhotic events and mortality of patients in two arms will be compared. The cutoff values of vPPG to spare endoscopies with low missed VNT (varices needing treatment) are preliminarily determined with the cohort data.

ELIGIBILITY:
Inclusion Criteria:

Inpatients (Shanghai Tongji Hospital) with cirrhosis, which is confirmed by the imaging tests (upper abdominal ultrasound/CT/MRI) or liver biopsy pathology.

Exclusion Criteria:

* 1. Portal vein embolism;
* 2. Splenectomy;
* 3. Hepatic encephalopathy;
* 4. Hepatic space occupying lesions (such as hepatic cysts, hemangiomas, etc.) with diameter > 3cm and local compression effect;
* 5. Contraindications of enhanced CT test, such as iodine allergy, peripheral veins are too thin to inject contrast medium;
* 6. Contraindications of upper GI endoscopy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed cirrhosis by imaging tests (upper abdominal ultrasound/CT /MRI) or liver biopsy pathology
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
The morbidity of cirrhotic decompensated events | 2 years
  The occurence rate of cirrhotic decompensated events of enrolled patients
The mortality of cirrhosis | 2 years
  Patients who die because of cirrhosis

SECONDARY OUTCOMES:
Spared endoscopies | 2 years
  Patients who don't need upper endoscopic monitoring
Number of missed VNT | 2 years
  Missed cases of patients who have varices needing treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tongji Hospital, Tongji University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No